CLINICAL TRIAL: NCT05134350
Title: A Phase 1, Open Label, Randomized, 2-Way Crossover, 3-Period Study to Evaluate the Effect of Food and a Proton Pump Inhibitor on the Pharmacokinetics of LOXO-305 in Healthy Adult Subjects
Brief Title: Study of the Effect of Food and a Proton Pump Inhibitor (PPI; Omeprazole) on LOXO-305 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-BTK-20014; J2N-OX-JZNH (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-10-22; First posted 2021-11-24 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — pirtobrutinib; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1: ABC (Experimental): * Period 1: Single oral dose of 200 milligram (mg) LOXO-305 (Fasted state) on Day 1 (Treatment A)
  * Period 2: Single oral dose of 200 mg LOXO-305 (Fed state) on Day 8 (Treatment B)
  * Period 3: Single oral dose of 40 mg Omeprazole (Fasted state) on Day 15 to 17 and single oral dose of 200 mg LOXO-305 + 40 mg Omeprazole (Fasted state) on Day 18 (Treatment C)
  A washout period of 7 days was maintained between each treatment period.
  Interventions: Drug: LOXO-305; Drug: Omeprazole
- Treatment Sequence 2: BAC (Experimental): * Period 1: Single oral dose of 200 mg LOXO-305 (Fed state) on Day 1 (Treatment B)
  * Period 2: Single oral dose of 200 mg LOXO-305 (Fasted state) on Day 8 (Treatment A)
  * Period 3: Single oral dose of 40 mg Omeprazole (Fasted state) on Day 15 to 17 and single oral dose of 200 mg LOXO-305 + 40 mg Omeprazole (Fasted state) on Day 18 (Treatment C)
  A washout period of 7 days was maintained between each treatment period.
  Interventions: Drug: LOXO-305; Drug: Omeprazole

INTERVENTIONS:
Drug: LOXO-305 — LOXO-305 orally.
Drug: Omeprazole — Omeprazole Orally.

SUMMARY:
The main purpose of this study is to learn about how food and a PPI (omeprazole) affect LOXO-305 in healthy participants. Participation could last about nine weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of non-childbearing potential.
* Within body mass index (BMI) range 18.0 to 32.0 kilograms per square meter (kg/m²).
* Participants will be in good general health, based on medical history, physical examination findings, vital signs, 12 lead electrocardiogram (ECG), or clinical laboratory tests, as determined by the Investigator (or designee).
* Able to comply with all study procedures, including the 25-night stay at the Clinical Research Unit and follow-up phone call.

Exclusion Criteria:

* History or presence of any of the following, deemed clinically significant by the Investigator (or designee), and/or Sponsor:

  * liver disease
  * pancreatitis
  * peptic ulcer disease
  * intestinal malabsorption
  * gastric reduction surgery
  * history or presence of clinically significant cardiovascular disease.
* Participants with out-of-range, at-rest vital signs.
* Abnormal laboratory values determined to be clinically significant by the Investigator (or designee), and Sponsor.
* Clinically significant abnormality, as determined by the Investigator (or designee), from physical examination.
* Participation in any other investigational study drug trial involving administration of any investigational drug in the past 30 days or 5 half-lives, whichever was longer, prior to the first dose administration (Day 1).
* Use or intention to use any prescription or over-the-counter medications within 14 days prior to the first dose administration (Day 1) through the end of the trial.
* History or presence, upon clinical evaluation, of any illness that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results, or put the participant at undue risk.
* Donation of blood from 56 days prior to Screening, plasma or platelets from 4 weeks prior to Screening.
* Receipt of blood products within 2 months prior to Check-in (Day -1).
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, biliary, renal, hematological, pulmonary, cardiovascular (including any prior history of cardiomyopathy or cardiac failure), GI, neurological, or psychiatric disorder (as determined by the Investigator), or cancer within the past 5 years (except localized basal cell, squamous, or in situ cancer of the skin).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renée Ward, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to 2 treatment sequences (ABC and BAC), with each sequence having 3 periods where participants were crossed over between the periods in each sequence. A washout period of 7 days was maintained between each treatment period.
Period: Period 1
Arm/Group | Treatment Sequence 1: ABC | Treatment Sequence 2: BAC
Started | 5 | 5
Received at Least 1 Dose of Study Drug | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Treatment Sequence 1: ABC | Treatment Sequence 2: BAC
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Period 3
Arm/Group | Treatment Sequence 1: ABC | Treatment Sequence 2: BAC
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Treatment Sequence 1: ABC: * Period 1: Single oral dose of 200 mg LOXO-305 (Fasted state) on Day 1 (Treatment A)
  * Period 2: Single oral dose of 200 mg LOXO-305 (Fed state) on Day 8 (Treatment B)
  * Period 3: Single oral dose of 40 mg Omeprazole (Fasted state) on Day 15 to 17 and single oral dose of 200 mg LOXO-305 + 40 mg Omeprazole (Fasted state) on Day 18 (Treatment C)
  A washout period of 7 days was maintained between each treatment period.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1: ABC | Treatment Sequence 2: BAC | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (10.66) | 35.2 (4.87) | 39.2 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve From Hour 0 to 24 (AUC [0-24]) Hours of LOXO-305
Description: PK: AUC(0-24) hours of LOXO-305 is reported. AUC(0-24) was calculated by the linear trapezoidal method.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post LOXO-305 dose
Population: All participants who received at least one dose of LOXO-305 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per milliliter
Groups:
- Treatment A: 200 mg LOXO-305 (Fasted): All the participants who received single oral dose of 200 mg LOXO-305 in fasted state on Day 1 (sequence 1), Day 8 (sequence 2).
- Treatment B: 200 mg LOXO-305 (Fed): All the participants who received single oral dose of 200 mg LOXO-305 in fed state on Day 1 (sequence 2), Day 8 (sequence 1).
- Treatment C: 200 mg LOXO-305 + 40 mg Omeprazole (Fasted): All participants in sequence 1 and 2 who received single oral dose of 40 mg Omeprazole in fasted state on Day 15 to 17 and single oral dose of 200 mg LOXO-305 + 40 mg Omeprazole in fasted state on Day 18.
Arm/Group | Treatment A: 200 mg LOXO-305 (Fasted) | Treatment B: 200 mg LOXO-305 (Fed) | Treatment C: 200 mg LOXO-305 + 40 mg Omeprazole (Fasted)
Number analyzed (Participants) | 10 | 10 | 10
hour*nanograms per milliliter | 55100 (17.5) | 51900 (12.8) | 59900 (15.5)

2. Primary Outcome: PK: Area Under the Concentration-time Curve From Hour 0 to the Last Measurable Concentration (AUC[0-t]) of LOXO-305
Description: PK: AUC(0-t) of LOXO-305 is reported. AUC(0-t) was calculated by linear trapezoidal method.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post LOXO-305 dose
Population: All participants who received at least one dose of LOXO-305 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per milliliter
Arm/Group | Treatment A: 200 mg LOXO-305 (Fasted) | Treatment B: 200 mg LOXO-305 (Fed) | Treatment C: 200 mg LOXO-305 + 40 mg Omeprazole (Fasted)
Number analyzed (Participants) | 10 | 10 | 10
hour*nanograms per milliliter | 89400 (17.8) | 85100 (19.3) | 99600 (17.1)

3. Primary Outcome: PK: Area Under the Concentration-time Curve Extrapolated to Infinity (AUC[0-Inf]) of LOXO-305
Description: PK: AUC(0-inf) of LOXO-305 is reported. AUC(0-inf) was calculated using the formula: AUC(0-inf) = AUC(0-t) + Ct/λZ; where Ct is the last measurable concentration and λZ is the apparent terminal elimination rate constant.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post LOXO-305 dose
Population: All participants who received at least one dose of LOXO-305 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per milliliter
Arm/Group | Treatment A: 200 mg LOXO-305 (Fasted) | Treatment B: 200 mg LOXO-305 (Fed) | Treatment C: 200 mg LOXO-305 + 40 mg Omeprazole (Fasted)
Number analyzed (Participants) | 10 | 10 | 10
hour*nanograms per milliliter | 90200 (17.6) | 86100 (18.9) | 101000 (16.8)

4. Primary Outcome: PK: Percentage Extrapolation for AUC0-Inf (%AUCextrap) of LOXO-305
Description: PK: %AUCextrap of LOXO-305 is reported.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post LOXO-305 dose
Population: All participants who received at least one dose of LOXO-305 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of extrapolation
Arm/Group | Treatment A: 200 mg LOXO-305 (Fasted) | Treatment B: 200 mg LOXO-305 (Fed) | Treatment C: 200 mg LOXO-305 + 40 mg Omeprazole (Fasted)
Number analyzed (Participants) | 10 | 10 | 10
percentage of extrapolation | 0.911 (27.2) | 1.12 (42.6) | 0.893 (34.5)

5. Primary Outcome: PK: Maximum Observed Plasma Concentration (Cmax) of LOXO-305
Description: PK: Cmax of LOXO-305 is reported.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post LOXO-305 dose
Population: All participants who received at least one dose of LOXO-305 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Treatment A: 200 mg LOXO-305 (Fasted) | Treatment B: 200 mg LOXO-305 (Fed) | Treatment C: 200 mg LOXO-305 + 40 mg Omeprazole (Fasted)
Number analyzed (Participants) | 10 | 10 | 10
nanograms per milliliter | 5450 (31.7) | 4340 (16.6) | 5490 (16.7)

6. Primary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of LOXO-305
Description: PK: tmax of LOXO-305 is reported.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post LOXO-305 dose
Population: All participants who received at least one dose of LOXO-305 and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: 200 mg LOXO-305 (Fasted) | Treatment B: 200 mg LOXO-305 (Fed) | Treatment C: 200 mg LOXO-305 + 40 mg Omeprazole (Fasted)
Number analyzed (Participants) | 10 | 10 | 10
hours | 2.50 [1.50 to 4.00] | 3.00 [1.00 to 4.00] | 2.25 [1.50 to 3.00]

7. Primary Outcome: PK: Apparent Terminal Elimination Half-life (t½) of LOXO-305
Description: PK: t½ of LOXO-305 is reported.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post LOXO-305 dose
Population: All participants who received at least one dose of LOXO-305 and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A: 200 mg LOXO-305 (Fasted) | Treatment B: 200 mg LOXO-305 (Fed) | Treatment C: 200 mg LOXO-305 + 40 mg Omeprazole (Fasted)
Number analyzed (Participants) | 10 | 10 | 10
hours | 20.2 (4.24) | 21.5 (5.75) | 19.7 (2.87)

8. Primary Outcome: PK: Apparent Systemic Clearance (CL/F) of LOXO-305
Description: PK: CL/F of LOXO-305 is reported.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post LOXO-305 dose
Population: All participants who received at least one dose of LOXO-305 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per Hours (L/h)
Arm/Group | Treatment A: 200 mg LOXO-305 (Fasted) | Treatment B: 200 mg LOXO-305 (Fed) | Treatment C: 200 mg LOXO-305 + 40 mg Omeprazole (Fasted)
Number analyzed (Participants) | 10 | 10 | 10
Liter per Hours (L/h) | 2.22 (17.6) | 2.32 (18.9) | 1.99 (16.8)

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 32
Description: All participants who received at least 1 dose of study drug.
Groups:
- Treatment C: 40 mg Omeprazole (Fasted): All participants who received single oral dose of 40 mg Omeprazole (Fasted) on Day 15 to 17.
Arm/Group | Treatment A: 200 mg LOXO-305 (Fasted) | Treatment B: 200 mg LOXO-305 (Fed) | Treatment C: 200 mg LOXO-305 + 40 mg Omeprazole (Fasted) | Treatment C: 40 mg Omeprazole (Fasted)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: 200 mg LOXO-305 (Fasted) (N=10) | Treatment B: 200 mg LOXO-305 (Fed) (N=10) | Treatment C: 200 mg LOXO-305 + 40 mg Omeprazole (Fasted) (N=10) | Treatment C: 40 mg Omeprazole (Fasted) (N=10)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT05134350/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT05134350/SAP_001.pdf